CLINICAL TRIAL: NCT00006203
Title: Naltrexone, Craving, and Drinking: Ecological Assessment
Brief Title: Naltrexone, Craving, and Drinking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Peter Monti, professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAAMON0785011A1; R01AA007850 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2006-10

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: After a one-week placebo lead-in period, drinkers were randomized to 3 weeks of daily naltrexone or placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone Arm (Experimental): Three weeks of daily 50mg Naltrexone
  Interventions: Drug: Naltrexone 50 Mg
- Placebo Arm (Placebo Comparator): Three weeks of daily placebo (sugar)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone 50 Mg — Daily 50 mg for 3 weeks
  Arms: Naltrexone Arm
Drug: Placebo — Daily doses of placebo for 3 weeks
  Arms: Placebo Arm

SUMMARY:
This 5-week study will examine the effects of naltrexone on alcohol craving, drinking rates, and reaction to drinking-related triggers, or cues, in participants' everyday environment and in laboratory sessions. Participants will monitor and record their daily desires to drink, environmental circumstances in which urges occur, and drinking behavior using a palm top computer. Participants will receive naltrexone or a placebo. One week after receiving medication, all participants will be asked to respond to alcohol-related cues that may or may not arouse the desire to drink.

ELIGIBILITY:
Inclusion Criteria:

* Drink at least 4 days per week with 2 heavy drinking days (more than 6 standard drinks for men, more than 5 drinks for women) per week on average during the month prior to the study.

Exclusion Criteria:

* Current interest in treatment or a history of treatment for alcohol problems.
* History of liver disease or current liver function tests greater than five times normal.
* Opiate abuse or dependence, any opiate use two weeks before the study or a urine test screen that is positive for opiates.
* Females, who are pregnant, nursing, or not using reliable birth control method.
* Daily use of acetaminophen.
* Living with someone who participated in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island, United States